CLINICAL TRIAL: NCT04222322
Title: The Effect of Epitomee Capsule on Body Weight in Patients With Overweight and Obesity With and Without Prediabetes
Brief Title: The Effect of Epitomee Capsule on Body Weight in Patients With Overweight and Obesity
Acronym: RESET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epitomee medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRT-05-031
Record Dates: First submitted 2019-12-30; First posted 2020-01-09 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Epitomee Capsule (Experimental): Epitomee Capsule combined with moderate intensity lifestyle counseling
  Interventions: Device: Epitomee Capsule
- Control-Placebo (Placebo Comparator): Visually matching (to Epitomee capsule) placebo capsule combined with moderate intensity lifestyle counseling
  Interventions: Other: Control-Placebo

INTERVENTIONS:
Device: Epitomee Capsule — Arm treatment: Epitomee Capsule combined with moderate intensity lifestyle counseling.
  Arms: Epitomee Capsule
Other: Control-Placebo — Arm treatment: Visually matching placebo capsule combined with moderate intensity lifestyle counseling.
  Arms: Control-Placebo

SUMMARY:
The effect of Epitomee Capsule on body weight in patients with overweight and obesity with and without Prediabetes

DETAILED DESCRIPTION:
This is a Prospective, Randomized, Double-blind, Placebo controlled, Multi-center, Pivotal, Adaptive trial designed to demonstrate that the use of Epitomee Capsule, in combination with lifestyle modification, is superior to the placebo device in reducing body weight at 24-weeks

ELIGIBILITY:
Inclusion Criteria:

1. Men or women >= 18 years
2. Current BMI of 25.0-40.0 kg/m2 inclusive
3. Eligible female subjects will be:

   Non-pregnant, evidenced by a negative urine dipstick pregnancy test Non-lactating Females will be either surgically sterile or postmenopausal or agree to continue using an accepted method of birth control during the study.
4. Normoglycemic subjects with both:

   1. Fasting plasma glucose <100 mg/dL
   2. HbA1c <5.7% or:

   Prediabetic subjects with either one or both of the following criteria:
   1. FPG≥100 mg/dL and <126 mg/dL
   2. 5.7% ≤ HbA1c ≤6.4% Naive Prediabetes or treated with metformin (up to 2000mg/dL inclusive)
5. Ability to provide informed consent before any trial-related activities
6. Ability and willingness to complete the physical activity in accordance to the study's exercise program
7. Willingness to maintain a diet in accordance with study requirement for the duration of the study
8. Subjects must have:

   * A primary care provider who is responsible for providing routine care
   * A reliable telephone or internet service to communicate with study staff
9. Understand and be willing to comply with all study-related procedures and agree to participate in the study by giving written informed consent
10. Study subjects must be willing to notify the staff of any change in their medical health (including surgeries) or change in drug treatments (addition of drugs, stopping of drugs, or change in drug dose) during the course of the trial.
11. Previously attempted to lose weight unsuccessfully using a medically supervised or self-directed diet.
12. Willingness to avoid medications or other substances known to affect weight changes during the study
13. Willingness to avoid non-steroidal anti-inflammatory drugs (NSAIDs) other than low dose aspirin including Diclofenac, Ibuprofen, Naproxen, or other medications known to be gastric irritants during the study.
14. Subjects on psychiatric medications are clinically well-controlled with a stable psychiatric medication dose for at least 3 months prior to study entry.

Exclusion Criteria:

1. Pregnant or nursing, or plans to become pregnant in the next 12 months, or not using adequate contraceptive measures
2. Weight loss of more than 10 pounds in the past 6 months
3. Use in the past 6 months of medications or other substances known to induce weight gain or weight loss
4. Participation in any clinical study (weight-loss or non-weight loss study) within the past 3 months
5. Known history of endocrine disorders affecting weight, such as uncontrolled abnormal thyroid function, hypothalamic tumors, Cushing's syndrome, or other genetic syndromes
6. Currently receiving chronic steroid or immunosuppressive therapy
7. Subjects previously diagnosed with HIV, hepatitis B or C
8. Subjects diagnosed with bulimia, binge eating disorder, compulsive overeating, high liquid calorie intake, or similar eating related psychological disorders
9. Intent to undergo gastric surgery or gastric banding during the study period or within the 6-month period after completion of this study
10. Prior use of any weight loss gastric medical device such as gastric balloon or gastric aspiration device
11. Known history of structural or functional disorders of the esophagus that may impede passage of the device through the gastrointestinal tract, including: Barrett's esophagus, esophagitis, dysphagia, achalasia, stricture/stenosis, esophageal varices, esophageal diverticula, esophageal perforation, or any other disorder of the esophagus
12. Known history of any swallowing disorder, esophageal chest pain disorders, or drug refractory esophageal reflux symptoms
13. Known history of structural or functional disorders of the stomach including, gastric ulcer, chronic gastritis, gastric varices, hiatal hernia (> 2 cm), cancer or any other disorder of the stomach or any symptoms of chronic upper abdominal pain, chronic nausea, chronic vomiting, chronic dyspepsia or symptoms suggestive of gastroparesis, including post-prandial fullness or pain, post-prandial nausea or vomiting or early satiety.
14. Known history of duodenal ulcer, intestinal diverticula (diverticulitis), intestinal varices, intestinal stricture/stenosis, small bowel obstruction, or any other obstructive disorder of the gastrointestinal (GI) tract
15. Currently have ongoing symptoms suggestive of intermittent small bowel obstruction, such as recurrent bouts of post-prandial abdominal pain, nausea or vomiting
16. Known history of irritable bowel syndrome, radiation enteritis or other inflammatory bowel disease, such as Crohn's disease
17. Known history of GI surgeries that may have resulted in anatomical GI tract abnormalities such as a stoma, Nissen Fundoplication or narrowing of any portion of the digestive tract. Examples of these GI surgeries include, but are not limited to, gastric banding; however, uncomplicated appendectomies are acceptable. In addition, known history of any surgeries that may have resulted in anatomical GI tract abnormalities such intestinal adhesions, or any other condition that may inhibit passage through any portion of the GI tract must be excluded
18. Subjects with Type 1 diabetes or type 2 diabetes
19. Experienced a myocardial infarction, has a known history of angina, underwent coronary bypass, a known history of congestive heart failure, or is currently being medically treated for any other cardiac condition
20. Poorly controlled hypertension (≥ 160 mmHg systolic and ≥ 100mmHg diastolic)
21. End stage renal disease or requiring hemodialysis within the past 6 months
22. Subjects taking medications on specified hourly intervals that may be affected by changes to gastric emptying, such as anti-seizure or anti-arrhythmic medications
23. Subjects requiring the use of anti-platelet drugs (except for low dose Aspirin as mentioned above) or other agents affecting the normal clotting of blood
24. Study subjects must not have a history of substance use disorder (licit or illicit) drug or alcohol abuse/addiction within 5 years of visit #1 (i.e. day of signing the informed consent document).
25. Study subjects must not have a medical history of sensitivity, intolerance, or toxicity to the investigational product, or agents similar to the investigational product.
26. Study subjects must not have a history of anaphylaxis or anaphylactoid reaction to any prior drug or supplement of any kind.
27. Study subjects must not have a history of cancer with the exception of non-melanoma skin cancer and "in situ" cancer of the cervix.
28. Study subjects must not be anticipating a significant change in job, job duties, or job work hours, which might impair their ability and willingness to undergo study-related procedures under the timelines specified by protocol, and otherwise impede their completion of the study.
29. Study subjects must not anticipate a reasonable likelihood of moving away from the research site, wherein such a move might impair their ability and willingness to undergo study-related procedures within the timelines specified by protocol, or otherwise impede their completion of the study.
30. Subjects who stopped smoking within 6 months prior to Screening Visit or considering smoking cessation during the study
31. Subjects who are habitual laxative users or using prescription medication for chronic constipation
32. Study subjects must not have change in medications treating hypertension and/or dyslipidemia within 1 month prior to Screening Visit (including change in dose)
33. Life expectancy less than 1 year or severe renal, hepatic, pulmonary or other medical condition.
34. Subject is employed by the investigator, or is a close relative of the investigator, or the investigator's staff
35. Subject is a close relative of another subject already enrolled in the study or lives in the same home with another subject enrolled in the study.
36. Subjects on psychiatric medications with no lifetime history of suicidal behavior.
37. Any other condition that, in the opinion of the investigator, would interfere with subject participation, may confound the study results, or interfere with compliance with the study (e.g., psycho-social issues).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
The difference between the percent body weight loss between the active and control groups | 24 weeks
  The difference between the percent average body weight loss at 24-weeks post randomization between the active and control groups
The proportion of treatment responders in the active group | 24 weeks
  The proportion of treatment responders defined as subjects who have lost 5% or more of baseline weight at 24-weeks post randomization, among the active group

CONTACTS AND LOCATIONS:
Overall Officials: Yael Kenan, Dr, Study Director — Epitomee Medical, VP Clinical Affairs
Locations (9):
- United States (9):
  - University of Alabama, Dept of Nutrition Sciences, Birmingham, Alabama
  - Northwestern University - 645 N. Michigan Avenue, Suite 530, Chicago, Illinois
  - The University of Kansas, Department of Internal Medicine, Kansas City, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Pennington Biomedical Research Center , 6400 Perkins Road, Baton Rouge, Louisiana
  - Wake Forest School of Medicine, Wake Forest Baptist Health - 525 Vine Street, 5th Floor, Suite 5119, Winston-Salem, North Carolina
  - Center for Weight and Eating Disorders at Perelman School of Medicine University of Pennsylvania - 3400 Civic Center Boulevard, Building 421,, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Weight Management Center - 67 President Street, Suite 410 South, Charleston, South Carolina
  - Juno Resreach, Houston, Texas

REFERENCES:
- [Derived] Bays HE, Ard JD, O'Neil PM, Wadden TA, Kushner RF, Jakicic JM, Wyatt HR, Greenway FL, Kamar M, Ganon-Elazar E, Asaraf LC, Ryan DH. Weight and cardiometabolic effects of a novel oral shape-shifting superabsorbent hydrogel capsule: Prespecified and exploratory analysis of the Epitomee capsule RESET study. Obes Pillars. 2025 Jan 31;13:100163. doi: 10.1016/j.obpill.2025.100163. eCollection 2025 Mar. PMID 40028615